CLINICAL TRIAL: NCT05143931
Title: Evaluating Environmental Control (AVOID) and Inhibitory Control (RESIST) Strategies to Improve Weight Management Outcomes
Brief Title: Avoid and Resist Strategies for Weight Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: University of California, Riverside (Other); WW International Inc (Industry); The University of Tennessee, Knoxville (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Northeastern University (Other)
Responsible Party: Principal Investigator, Sarah Salvy, Professor, Department of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001652; 1R01DK130851-01 (NIH)
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: single-site, prospective, four-parallel-arm, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- WW Only (Active Comparator): WW is commercially-available weight management program focusing on diet, physical activity and mindset skills.
  Interventions: Behavioral: WW
- WW + Home modification and grocery delivery (AVOID) (Experimental): WW + modification of home food environment + online grocery shopping and delivery
  Interventions: Behavioral: Home food environment and grocery delivery (AVOID); Behavioral: WW
- WW + Inhibitory control training (RESIST) (Experimental): WW + daily gamified inhibitory control training
  Interventions: Behavioral: Inhibitory control training (RESIST); Behavioral: WW
- WW + Home food modification and grocery delivery (AVOID) + Inhibitory control training (RESIST) (Experimental): WW + modification of home food environment + online grocery shopping and delivery + daily gamified inhibitory control training
  Interventions: Behavioral: Home food environment and grocery delivery (AVOID); Behavioral: Inhibitory control training (RESIST); Behavioral: WW

INTERVENTIONS:
Behavioral: Home food environment and grocery delivery (AVOID) — Participants (Arms 2 & 4) will receive 6 months of coaching (Zoom and/or email/text) to modify their home food environment and alter cues to promote healthy food choices
  Arms: WW + Home food modification and grocery delivery (AVOID) + Inhibitory control training (RESIST); WW + Home modification and grocery delivery (AVOID)
Behavioral: Inhibitory control training (RESIST) — Participants assigned to RESIST (Arms 3 & 4) will receive 6 months of coaching (Zoom and/or email/text) and gamified inhibitory control training.
  Arms: WW + Home food modification and grocery delivery (AVOID) + Inhibitory control training (RESIST); WW + Inhibitory control training (RESIST)
Behavioral: WW — Participants assigned to all arms will receive 6 months of coaching (Zoom and/or email/text) and commercially-available weight management program focusing on diet, physical activity and mindset skills.

SUMMARY:
The proposed randomized controlled trial tests two self-regulatory approaches to improve intentional weight loss and diet quality in individuals with overweight or obesity: (1) an environmental control strategy (AVOID) and (2) an impulse control training strategy (RESIST).

DETAILED DESCRIPTION:
Evidence-based weight management programs are effective when individuals are able to consistently adhere to recommendations. However, a large proportion of treatment-seeking individuals do not experience clinically significant weight loss. Innovative strategies are needed to optimize behavior change in weight management interventions. The proposed randomized controlled trial tests two self-regulatory approaches to improve intentional weight loss and diet quality in individuals with overweight or obesity: (1) an environmental control strategy (AVOID) and (2) an impulse control training strategy (RESIST). Specifically, 500 women and men (BMI between 25-45 kg/m2) will be recruited from the Cedars-Sinai Medical Center network of hospitals and clinics. All participants will be enrolled in a 12-month weight-management program (WW, formerly Weight Watchers©) focusing on diet, physical activity and mindset skills, and randomized to one of four study arms: (1) WW only, (2) WW + modification of home food environment and online grocery delivery (AVOID), (3) WW + gamified inhibitory control training (RESIST), (4) WW + AVOID + RESIST. Baseline, 6- and 12-month assessments will be completed by experienced, English and Spanish speaking study staff. Aim 1 (Outcomes). (a) Tests how AVOID and RESIST affect weight loss and waist circumference (primary) and diet quality (secondary). H1a: AVOID and/or RESIST (arms 2, 3, 4) will result in greater weight loss at 6-month and 12-month timepoints compared to WW alone. (b) Tests potential ripple effects of AVOID and RESIST on available household members' diet quality (primary) and weight (secondary). H1b: The investigators predict that AVOID (arms 2 and 4) will produce greater dietary changes in household members than WW alone and RESIST (arms 1 and 3). Aim 2 (Mechanisms). Tests the mechanistic pathways of AVOID and RESIST by (a) comparing longitudinal changes in inhibitory control and home food environment across study arms; and (b) whether inhibitory control and the home food environment mediate the relationships between study arms and anthropometric and dietary outcomes. H2: AVOID will produce changes in the home food environment and RESIST will operate on inhibitory control. Aim 3 (Moderators). Examines how (a) individual characteristics (age, sex, ethnicity, socioeconomic status, household composition, physical activity, baseline BMI and executive functioning), and (b) process data (frequency of grocery delivery, dining out and take out, impulse control training and WW app use) moderate the relationship between study arms and anthropometric and dietary outcomes. These considerations are important to help explain heterogeneity in intervention outcomes and to understand who benefits from AVOID and/or RESIST.

ELIGIBILITY:
Inclusion Criteria (Main participants):

* Age 18 years or older
* BMI between 25-45 kg/m2
* Read, write, and speak English with acceptable visual acuity
* Has a household member (≥ 14 years) willing to complete three brief assessments over 12 months* *Only applies to individuals who indicate they are cohabitating with at least one eligible household member

Inclusion Criteria (Household participants):

* 14-years-old
* Parent consent for children <18-years-old
* Willingness to complete assessments / measurements

Exclusion Criteria (Main participants):

* Currently enrolled in weight loss interventions or undergoing bariatric surgery
* Pregnant women
* Individuals for whom weight loss may be contraindicated (e.g., unstable coronary artery disease, end-stage disease, active cancer treatment, uncontrolled insulin-dependent diabetes, portal hypertension, drug/alcohol abuse)
* Individuals with severe cognitive delays or visual/hearing impairment
* Individuals who are unable or unwilling to complete the study assessments / measurements

Exclusion Criteria (Household participants):

* ≤ 14-years-old
* Individuals who are unable or unwilling to complete the study assessments / measurements

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Change in BMI from baseline to 12 months. | Baseline, 6-month, 12-month
  BMI will be calculated by aggregating participants' self-reported height in meters and weight in kilograms at baseline, 6- and 12-months.

SECONDARY OUTCOMES:
Diet quality assessed by 24h-dietary recall | Baseline, 6-month, 12-month
  Gold standard interviewer-administered, multi-pass 24h-recalls (2 weekdays, 1 weekend day) will be used to measure diet quality. The Nutrition Data System for Research software (Nutrition Coordinating Center, University of Minnesota) is used to analyze the data. Investigators will use the 24h-recalls to assess changes in participants and household members' overall diet quality, based on adherence to the dietary guidelines for fruits and vegetables, servings of whole grains, red/processed meat, alcoholic beverages and food/beverages with added sugars.

OTHER OUTCOMES:
Home availability of healthy and unhealthy foods and beverages | Baseline, 6-month, 12-month
  Participants will self-report the availability of fruits and vegetables, servings of whole grains, red/processed meat, alcoholic beverages and food/beverages with added sugars in participants' homes. Responses will be scored as availability of healthy foods and beverages (e.g., fruits and vegetables), and availability of less healthy foods and beverages (e.g., processed meat, food/beverages with added sugars).
Flanker task | Baseline, 6-month, 12-month
  Participants have 1000ms to identify which direction a central arrow is pointing. Participants complete 64 congruent and incongruent randomly mixed trials. In congruent trials flanking stimuli points in the same direction as the central stimulus while in incongruent trials flanking stimuli points in the opposite direction.
Continuous Performance Task Go/No-Go | Baseline, 6-month, 12-month
  Participants respond to a target shape (e.g. a white five-pointed star) and withhold a response from non-target shapes. In 20% of presented trials an inhibitory response will be required.
Set-Shifting | Baseline, 6-month, 12-month
  Participants categorize colored shapes by color or shape in three blocks. In the first two blocks, participants categorize shapes for 20 trials. In the third block, the categorization rules are randomly interleaved, and participants switch between rules. Participants have 1500ms to identify the stimulus and complete 96 trials with a 25% chance of rule-switching.
Demographics | Baseline only
  Participants will complete a questionnaire surveying: date of birth, sex, socioeconomic status (education level, household income, marital status, employment status), household composition (multigenerational, single, married, cohabitating, children) and race/ethnicity.
Executive Functioning | Baseline, 6-month, 12-month
  The Behavior Rating Inventory of Executive Function®- Adult Version (BRIEF-A) is a standardized measure of executive functions or self-regulation in everyday environment. The BRIEF-A assesses nine non-overlapping theoretically and empirically derived clinical scales: Inhibit, Self-Monitor, Plan/Organize, Shift, Initiate, Task Monitor, Emotional Control, Working Memory, and Organization of Materials. BRIEF-A is available in English and Spanish and can be computer-administered. Baseline score on the BRIEF will be tested as moderator of the relationships between study arms and outcomes.
WW Process Data | monthly between baseline and 12-month
  Interactions such as tracked food, weight and activity in WW app will be passively recorded to operationalize engagement. A higher score indicates greater engagement.
Grocery Delivery Process data | monthly between baseline and 12-month
  Frequency of grocery delivery and dining out/take out will be recorded through participants' self-report of grocery delivery. Higher frequencies of grocery delivery indicates greater engagement.
PolyRules! Process data | monthly between baseline and 12-month
  Frequency/duration of gamified cognitive training will be passively recorded by the PolyRules! app. Greater frequency and duration indicate greater engagement.
Physical activity | Baseline, 6-month, 12-month
  The International Physical Activity Questionnaire (IPAQ) will be used to assess activity in 5 domains: job-related; transportation; housework, house maintenance, and caring for family; recreation, sport, and leisure-time physical activity; and time spent sitting. Data conferred by the WW program will also be leveraged, as participants track their activity (type, duration and intensity) via the WW mobile app or online website. Investigators will examine how engagement in exercise and daily activities moderate the relationships between study arms and outcomes.
Eating attitudes | Baseline, 6-month, 12-month
  The Dutch Eating Behavior Questionnaire (DEBQ) will be used to assess participants' approach to food and eating along three dimensions: emotional, external and restricted eating. There is a high degree of stability for each of these three eating behavior scales. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Food Security Questionnaire | Baseline only
  The Food Security Questionnaire will be used to evaluate the availability of nutritious and safe foods for participants and their households at all times. The questionnaire will assess the household's ability to meet their food needs and will determine their placement on a food security continuum based on their responses to a series of questions. Researchers will analyze how food security impacts the relationships between different study arms and the outcomes.
Changes in Health and Lifestyle. | 6-month, 12-month
  Changes in health, medication, diet, and exercise among participants will be assessed via routine questionnaires administered at specific study time points (e.g., 6 and 12 months). The study team will monitor reported changes on an ongoing basis. Any data indicating potential new exclusion criteria (e.g., a diagnosis of cancer or other serious conditions) will be reviewed on a case-by-case basis. If the data meet the criteria for New Reportable Information (NRI), such as adverse events or single-subject exemptions, the appropriate reporting procedures will be followed according to IRB guidelines.
Participant Experience Interview | withdrawal or 6-month and 12-month
  Main participants will be asked to complete a brief semi-structured participant experience interview at 6 months and at the conclusion of their intervention (either at withdrawal or 12-months). The interview will be conducted online via Zoom or MS Teams and last between 10-15 minutes. The questions asked will vary depending on the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah-Jeanne Salvy, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sobolev M, Ruiz J, Diniz MA, Raynor H, Foster GD, Seitz AR, Salvy SJ. Preference for behavior change strategies in randomized controlled trials: Evidence from weight management. Contemp Clin Trials. 2025 Sep;156:108031. doi: 10.1016/j.cct.2025.108031. Epub 2025 Jul 28. PMID 40738220
- [Derived] Caceres NA, Yu Q, Capaldi J, Diniz MA, Raynor H, Foster GD, Seitz AR, Salvy SJ. Evaluating environmental and inhibitory control strategies to improve outcomes in a widely available weight loss program. Contemp Clin Trials. 2022 Aug;119:106844. doi: 10.1016/j.cct.2022.106844. Epub 2022 Jul 5. PMID 35798248